CLINICAL TRIAL: NCT07210749
Title: A Phase II Trial Assessing 12 Gy in 6 Fractions Radiotherapy for Low-Grade B-cell Orbital Lymphoma
Brief Title: Radiotherapy 12Gy in 6 Fractions For Orbital Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Matthew Chan, Principal Investigator (Co-PI), British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-OLY
Record Dates: First submitted 2025-09-22; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Orbital Lymphoma
MeSH Terms: conditions — Orbital lymphoma

STUDY DESIGN:
Intervention Model Description: 12 Gy in 6 fractions external beam radiotherapy using standard-of-care radiation volumes for low-grade orbital lymphoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 Gy in 6 fractions of external beam radiation therapy (Experimental): 12 Gy in 6 fractions of conventional external beam radiation therapy using standard-of-care radiation volumes for low-grade orbital lymphoma
  Interventions: Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — 12 Gy in 6 fractions of external beam radiation therapy

SUMMARY:
Current standard RT doses (24-25Gy) provide excellent disease control for patients with indolent B-cell orbital lymphoma, but can cause significant late toxicities. Ultra-low dose RT (4Gy in 2 fractions) has minimal toxicity but lower disease control, requiring intensive follow-up to salvage persistent tumors. Some centers are moving towards this dose as the new standard. A recent study using 12Gy in 4 fractions to any body site showed early data suggesting high disease control rates with minimal toxicity. This study assesses 12Gy in 6 fractions, aiming to enhance disease control over 4Gy while reducing toxicity compared to 24Gy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with stage I-IV indolent NHL*
* Able to provide informed consent
* Histologically confirmed indolent NHL involving one or both orbits. If bilateral, biopsy of only one orbit is permitted as long as high clinical suspicion of contralateral orbit involvement
* Measurable orbital disease after biopsy, either clinically or radiographically
* ECOG performance status 0-3
* Life expectancy >12 months
* Available for treatment and follow-up (including scheduled post-treatment imaging and ophthalmologic exam)
* Able and willing to complete quality of life questionnaires via paper or online portal if they provide their email address on the informed consent document

  * Stage II-IV allowed but if systemic therapy given after RT the timing will be recorded, and subjects will be stratified according to receipt of systemic therapy

Exclusion Criteria:

* Aggressive NHL histology (including grade 3B follicular lymphoma)
* Prior RT to orbit
* Patients requiring treatments outside standard clinical hours
* Systemic therapy for lymphoma is not permitted within the period of time between 2 weeks prior to RT start and 2 weeks after RT completion
* Patients who are pregnant
* History of other malignancy within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death and/or treated with expected curative outcome (for example, appropriately treated non-melanoma skin cancer, carcinoma in-situ of the cervix, localized prostate cancer, breast ductal carcinoma in-situ, or stage I endometrial cancer)
* Any medical condition that, in the investigator's judgement, would preclude the individual's safe participation in and completion of the study, or could affect interpretation of the results (e.g. pre-existing retinopathy, active connective tissue disease)
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2035-08-31 (Estimated); Study Completion 2036-08-31 (Estimated)

PRIMARY OUTCOMES:
Assess 2-year orbital LC after 12 Gy in 6 fractions. | 24 Months after Treatment

SECONDARY OUTCOMES:
Response rates (complete/partial/minimal response, stable/progressive disease) | 6 months and 12 months after treatment
Evaluate orbital local control | 5 years after treatment
Assess freedom from further in-field RT (FFRT), freedom from distant relapse (FFDR) and overall survival (OS) | 2 year and 5 year after treatment
Health-Related Quality of Life using the EORTC QLQ-C30 | 5 years after treatment
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) measures health-related quality of life through 5 functional, 9 symptom, and 1 global health status scale; minimum score = 0, maximum score = 100 (for functional scales, higher is better; for symptom scales, lower is better)
Ocular Toxicity per CTCAE (5.0) | 2 year and 5 year after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Vancouver, Vancouver, British Columbia, Canada